CLINICAL TRIAL: NCT03530527
Title: Endoscopic Retrograde Cholangiopancreatography Versus Endoscopic Ultrasound Guided Biliary Drainage in Inoperable Malignant Distal Bile Duct Obstruction
Brief Title: Endoscopic Biliary Drainage in Malignant High Grade Biliary Stricture
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated because of difficulty in completing the study as originally planned
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Nisa Netinatsunton, Secretory of NKC Institute of Gastroenterology and Hepatology, Prince of Songkla University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC 60-277-21-1
Record Dates: First submitted 2018-05-08; First posted 2018-05-21 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Malignant Biliary Stricture
Keywords: ERCP; Endoscopic ultrasound (EUS) guided biliary drainage
MeSH Terms: interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ERCP with biliary stenting (Active Comparator): Patient will be undergone ERCP with biliary stenting for biliary decompression to relieve biliary obstruction.
  Interventions: Procedure: ERCP with biliary stenting
- EUS guided biliary drainage (Active Comparator): Patient will be undergone EGBD for biliary decompression to relieve biliary obstruction.
  Interventions: Procedure: EUS guided biliary drainage

INTERVENTIONS:
Procedure: ERCP with biliary stenting — ERCP with biliary stent is performed using a side view duodenoscope of Olympus (TJF-160). Biliary cannulation is performed using a sphincterotome and 0.035 inch jag wire, and cholangiogarm is done to assess common bile duct diameter, and length of biliary stricture. Biliary sphincterotomy is then performed. A straight biliary stent is placed across stricture bile duct.
  Other Names: G1
  Arms: ERCP with biliary stenting
Procedure: EUS guided biliary drainage — EUS guided biliary drainage is performed using a linear echoendoscope of Olympus (GFUCT240). Extrahepatic bile duct was identified from duodenal bulb, then 19 G needle is inserted into bile duct with confirmed with cholangiogram. The fistula tract is dilated using a 6 Fr cystotome (Wilson Cook Medical). A double pigtail stent is placed across biliary-enteric fistula.
  Other Names: G2
  Arms: EUS guided biliary drainage

SUMMARY:
Biliary drainage is the mainstay of the palliative treatment in patients with inoperable malignant bile duct stricture. Endoscopic retrograde cholangiopancreatography (ERCP) is the cornerstone of biliary drainage method in these patients. However, ERCP is sometime unsuccessful to perform because of the presence of the high grade biliary stricture, tumor invasion of duodenum and ampulla of vater and surgically altered gastrointestinal anatomy. Endoscopic ultrasound (EUS) guided biliary drainage has been emerged as an alternative procedure to traditional surgical bypass and percutaneous trans hepatic biliary drainage after failed ERCP. There were few data to directly compare between ERCP and EUS guided biliary drainage and in patients with malignant high grade biliary stricture.

DETAILED DESCRIPTION:
The aim of this study is comparing the efficacy and complications between ERCP and EUS guided biliary drainage in patients with malignant high grade biliary stricture. Malignant high grade biliary stricture has not been well defined. The investigators define this malignant high grade biliary stricture using these arbitrary number include total bilirubin ≥ 15 mg/dl and or bile duct diameter ≥12 mm. based on the investigation's experience.

The study will be divided patients with inoperable malignant high grade biliary stricture into 2 groups, group (A) will be undergone ERCP with biliary stenting and group (B) will be undergone EUS guided biliary drainage. If the assigned intervention is not successful, then patients will be crossed-over to the another intervention.

ELIGIBILITY:
Inclusion Criteria: I) Patients aged > 18 years. II) Clinical, laboratory data, imaging and or histology suggestive of malignant distal bile duct strictures that occurs as a result of pancreatic adenocarcinoma, cholangiocarcinoma, ampullary carcinoma, duodenal carcinoma, gallbladder cancer and metastasis malignant bile duct obstruction III) Inoperability by tumor staging, medically unfit or patient wishes

1. distant metastasis
2. major vascular involvement (unreconstructible Superior mesenteric vein/Portal vein, superior mesenteric artery, common hepatic artery and celiac artery)
3. metastasis to lymphnode beyond the field or surgery IV) Jaundice, total bilirubin ≥15 mg/dl and/ or Common bile duct diameter ≥12 mm

Exclusion Criteria: I) pregnancy II) uncorrectable coagulopathy ( international normalized ratio ≥ 1.5 ) III) thrombocytopenia (platelet count < 50,000 ) IV) extremely poor general condition, ERCP with stent insertion impossible for ethical reasons V) an extension of stricture to the main biliary confluent (hilum) or the existence of obstructive duodenal invasion VI) active suppurative cholangitis VI) surgically altered anatomy (i.e. Billroth II or Roux-en-Y reconstruction ) VII ) previous treatment with bile duct stent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2018-11-28 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
Technical success rate | 24 hours
  The number of patients with success of placement of stent in the desired. location

SECONDARY OUTCOMES:
Clinical success rates | 2 weeks
  The number of patients with total bilirubin drop more than 30 % compare with baseline after successful biliary stent placement.
Total procedure time | 24 hours
  The time interval between the intubation of the scope until the placement of the stent
The complication rates | 4 weeks
  The number of patients who developed complications related procedure included pancreatitis, bleeding, perforation, cholangitis as defined and graded according to the consensus guideline.
The mortality rates | 1 weeks
  The number of patients with death related to the procedure.
Stent patency | 12 weeks
  The time interval between biliary stent insertion and the need for unscheduled re-interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Nisa Netinatsunton, MD., Principal Investigator — NKC Institute of Gastroenterology and Hepatology, Faculty of Medicine, Prince of Songkla University, Hatyai, Songkhla, Thailand, 90110.
Locations (2):
- Thailand (2):
  - NKC Institue of Gastroenterology and Hepatology, Prince of Songkla University, Hat Yai, Changwat Songkhla
  - Prince of Songkla University, Hat Yai, Changwat Songkhla

IPD SHARING:
Plan to Share IPD: No
The individual data of patients participating in the study are not available for public sharing since the investigators did not obtain the consent to share the data of patient.